CLINICAL TRIAL: NCT05243524
Title: Phase 2b Single Arm Study of Maveropepimut-S and Low-Dose Cyclophosphamide in Subjects With Platinum-Resistant, Epithelial Ovarian Cancer.
Brief Title: Maveropepimut-S (MVP-S) and Low-Dose CPA in Patients With Platinum-Resistant Ovarian Cancer
Acronym: AVALON
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closure of IMV operations
Sponsor: ImmunoVaccine Technologies, Inc. (IMV Inc.) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1606-SUR-O25
Record Dates: First submitted 2022-02-07; First posted 2022-02-17 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Platinum-resistant Epithelial Ovarian Cancer
Keywords: T cell education; DPX-Survivac; Immunotherapy; Platinum-resistant (PROC); High grade serous (HGSOC)
MeSH Terms: interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MVP-S + CPA (Experimental): All subjects will receive two doses of maveropepimut-S (q3w) followed by up to six doses (q8w) plus low-dose cyclophosphamide on a repeating cycle of one week on/one week off.
  Interventions: Other: Maveropepimut-S; Drug: Cyclophosphamide 50mg

INTERVENTIONS:
Other: Maveropepimut-S — SC injection on days 7, 28, then q8w
  Other Names: MVP-S; DPX-Survivac
Drug: Cyclophosphamide 50mg — PO BID, one week on, one week off
  Other Names: CPA; Procytox; Cytoxan

SUMMARY:
Phase 2, single arm, study to assess the efficacy and safety of maveropepimut-S (MVP-S) and low-dose cyclophosphamide (CPA) in subjects with recurrent, platinum resistant ovarian cancer.

DETAILED DESCRIPTION:
A Simon two-stage statistical design to assess MVP-S in combination with low dose CPA in platinum-resistant epithelial ovarian cancer patients who have received no greater than 4 previous lines of anti-cancer therapy.

MVP-S, previously called DPX-Survivac, was recently evaluated in a small Phase 2 single arm study of ovarian cancer patients known as DeCidE1 (NCT02785250).

ELIGIBILITY:
Key Inclusion Criteria:

* Stage III or IV epithelial ovarian, fallopian tube, or primary peritoneal cancer, histologically diagnosed high-grade serous
* Platinum-resistant disease (relapsing within 3-6 months after completion of initial platinum-based treatment). Patients progressing at any time on or after ≥ 2nd platinum-based therapy are eligible.
* Received ≤ 4 prior lines of anti-cancer therapy for ovarian cancer, including at least one platinum-based therapy
* Evidence of progressive disease
* Measurable disease (RECIST v1.1) with at least one non-target lesion accessible by image-guided biopsy. No single lesion may be larger than 4 cm in diameter.
* Completed pre-treatment tumor biopsy and willing to undergo on-treatment tumor biopsy
* ECOG 0-1
* Live expectancy ≥ 6 months
* Meet protocol-specified laboratory requirements

Key Exclusion Criteria:

* Concurrent chemotherapy drugs, anti-cancer therapy or anti-neoplastic hormonal therapy, or radiotherapy
* Prior receipt of survivin-based vaccines/therapy, immune checkpoint inhibitors, IDO inhibitor, or cell-based therapy
* Non-epithelial tumor origin of the ovary, fallopian tube, or peritoneum
* Clinical ascites
* Concurrent second malignancy other than basal or squamous cell skin cancer, cervical carcinoma in situ, or Stage I or II caner in complete remission
* GI condition that might limit absorption of oral agents
* Recent history of thyroiditis
* History of autoimmune disease requiring treatment within the last two years (except paraneoplastic syndrome, vitiligo, or diabetes)
* History of bowel obstruction related to the disease
* Presence of a serious acute infection or chronic infection
* Uncontrolled concurrent illness or history of significant cardiac or pulmonary disfunction
* Myocardial infarction or cerebrovascular event within past 6 months
* Known central nervous system (CNS) or leptomeningeal metastasis (brain metastases)
* Clinically significant illness or major surgery within past 28 days or anticipated need for major surgery during study treatment
* Ongoing treatment with steroid therapy or other immunosuppressive
* Receipt of live attenuated vaccines
* Edema or lymphedema in the lower limbs > grade 2
* Acute or chronic skin and/or microvascular disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 13 months
  per RECIST v1.1 criteria

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 13 months
  per iRECIST criteria
Duration of Response (DOR) | up to 23 months
Disease Control Rate (DCR) | up to 13 months
Time to Progression (TTP) | up to 23 months
Progression Free Survival (PFS) | up to 23 months
Progression Free Survival (6m PFS) | at 6 months
Overall Survival (OS) | up to 23 months
CA-125 Response | up to 13 months
  monthly measurements
Frequency of adverse events | up to 13 months
  graded using NCI CTCAE v5.0

OTHER OUTCOMES:
Cell mediated immune response | up to 13 months
  analysis of PBMC/plasma samples
Changes in Tumor Micro-environment (TME) | up to 2 months
  analysis of paired biopsies

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - Stanford Health Care, Palo Alto, California
  - Ocala Oncology, Ocala, Florida
  - NYU Langone Hospital-Long Island, Mineola, New York
  - NYU Langone: Laura and Isaac Perlmutter Cancer Center, New York, New York
- CHUM - Centre hospitalier de l'Université de Montréal, Montreal, Quebec, Canada
- PanOncology Trials, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No